CLINICAL TRIAL: NCT00737672
Title: GORE VIABAHN® Endoprosthesis Versus Percutaneous Transluminal Angioplasty (PTA) to Revise Arteriovenous Grafts at the Venous Anastomosis in Hemodialysis Patients
Brief Title: GORE VIABAHN Endoprosthesis Versus Percutaneous Transluminal Angioplasty (PTA) to Revise AV Grafts in Hemodialysis
Acronym: REVISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVR 06-01; G070069 (Other: FDA (IDE))
Record Dates: First submitted 2008-08-15; First posted 2008-08-19 (Estimated); Results first posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Renal Failure; Hemodialysis
Keywords: Hemodialysis; Stent Graft; Venous Anastomosis; Arteriovenous Grafts
MeSH Terms: conditions — Renal Insufficiency | interventions — Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VIABAHN Treatment Group (Experimental): Use of GORE VIABAHN Endoprosthesis with PROPATEN Bioactive Surface to revise arteriovenous (AV) prosthetic grafts at the venous anastomosis in the maintenance or re-establishment of vascular access for hemodialysis as compared to Comparator Arm
  Interventions: Device: GORE VIABAHN Endoprosthesis with PROPATEN Bioactive Surface
- PTA Treatment Group (Active Comparator): Percutaneous Transluminal Angioplasty (PTA) in arteriovenous (AV) prosthetic grafts at the venous anastomosis in the maintenance or re-establishment of vascular access for hemodialysis as compared to Experimental Arm
  Interventions: Procedure: Percutaneous Transluminal Angioplasty

INTERVENTIONS:
Device: GORE VIABAHN Endoprosthesis with PROPATEN Bioactive Surface — Deployment of investigational stent graft at the venous anastomosis
  Arms: VIABAHN Treatment Group
Procedure: Percutaneous Transluminal Angioplasty — Percutaneous Transluminal Angioplasty at the venous anastomosis
  Arms: PTA Treatment Group

SUMMARY:
The objective of the study is to establish efficacy and safety of the GORE VIABAHN® Endoprosthesis with PROPATEN Bioactive Surface when used to revise arteriovenous (AV) prosthetic grafts at the venous anastomosis in the maintenance or re-establishment of vascular access for hemodialysis.

DETAILED DESCRIPTION:
The primary effectiveness hypothesis is to demonstrate that the GORE VIABAHN® Endoprosthesis with PROPATEN Bioactive Surface will extend the period of target lesion primary patency as compared to PTA.

The primary safety hypothesis is to demonstrate that the proportion of subjects remaining free from major device, procedure, and treatment site-related adverse events through 30 days post-procedure in the GORE® VIABAHN® Device group is not inferior to that of the PTA group.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patient with a dysfunctional or thrombosed forearm or upper arm prosthetic vascular access graft.
* The target lesion starts less than or equal to 30 mm from the venous anastomosis.
* The target lesion has > 50% stenosis as measured per protocol.
* The patient has a maximum of one secondary stenosis.

Exclusion Criteria:

* The age of the hemodialysis access graft is less than or equal to 30 days old from the date of the study procedure.
* The patient has undergone an intervention (surgical or percutaneous) of the vascular access circuit less than or equal to 30 days from the date of the study procedure.
* The secondary lesion is an occlusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2008-09; Primary Completion 2011-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Vesely, MD, Study Director — Vascular Access Center; Frontenac, MO
Locations (29):
- United States (29):
  - Birmingham, Alabama
  - Fresno, California
  - Inglewood, California
  - Oceanside, California
  - Riverside, California
  - San Diego, California
  - San Francisco, California
  - New Haven, Connecticut
  - Jacksonville, Florida
  - Albany, Georgia
  - Chicago, Illinois
  - Des Moines, Iowa
  - Louisville, Kentucky
  - Baltimore, Maryland
  - New Brighton, Minnesota
  - Saint Paul, Minnesota
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Greenville, South Carolina
  - Beaumont, Texas
  - Houston, Texas
  - Norfolk, Virginia
  - Winchester, Virginia
  - Bellevue, Washington
  - Spokane, Washington
  - Milwaukee, Wisconsin

REFERENCES:
- [Derived] Mohr BA, Sheen AL, Roy-Chaudhury P, Schultz SR, Aruny JE; REVISE Investigators. Clinical and Economic Benefits of Stent Grafts in Dysfunctional and Thrombosed Hemodialysis Access Graft Circuits in the REVISE Randomized Trial. J Vasc Interv Radiol. 2019 Feb;30(2):203-211.e4. doi: 10.1016/j.jvir.2018.12.006. PMID 30717951

RESULTS

PARTICIPANT FLOW:
Groups:
- PTA Treatment Group: Percutaneous Transluminal Angioplasty (PTA)in arteriovenous (AV) prosthetic grafts at the venous anastomosis in the maintenance or re-establishment of vascular access for hemodialysis as compared to Experimental Arm
  Percutaneous Transluminal Angioplasty: Percutaneous Transluminal Angioplasty at the venous anastomosis
Period: Overall Study
Arm/Group | VIABAHN Treatment Group | PTA Treatment Group
Started | 145 | 148
Exclusions Due to Protocol Deviations | 14 | 10
Per Protocol Population | 131 | 138
Completed | 65 | 65
Not Completed | 80 | 83
Not completed — Graft Abandonment | 48 | 56
Not completed — Death | 23 | 22
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Miscellaneous | 7 | 1
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VIABAHN Treatment Group | PTA Treatment Group | Total
Number analyzed (Participants) | 145 | 148 | 293
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.2 (12.9) | 61.3 (15.0) | 61.7 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 75 | 151
  Male | 69 | 73 | 142
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 30 | 46
  Not Hispanic or Latino | 126 | 114 | 240
  Unknown or Not Reported | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 9 | 7 | 16
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 74 | 80 | 154
  White | 61 | 56 | 117
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 4
Region of Enrollment [Number; unit: Participants]
  United States | 145 | 148 | 293
Body Mass Index [Mean (Standard Deviation); unit: Kg/m^2] | 29.7 (9.1) | 29.5 (8.6) | 29.6 (8.8)
History of Diabetes [Number; unit: Participants]
  History of Diabetes = YES | 94 (64.8) | 98 (66.2) | 192
  History of Diabetes = NO | 51 | 50 | 101
History of Hypertension [Number; unit: Participants]
  History of Hypertension = YES | 143 | 144 | 287
  History of Hypertension = NO | 2 | 4 | 6
Age of Vascular Access Graft [Mean (Standard Deviation); unit: Years] | 1.93 (1.92) | 2.28 (2.64) | 2.11 (2.31)
Total Number of Prior Interventions at the Target Lesions [Mean (Standard Deviation); unit: Number of Prior Interventions] | 1.85 (2.20) | 1.81 (2.34) | 1.83 (2.27)
Total Number of Prior Interventions to the Current Prosthetic Graft or Circuit [Mean (Standard Deviation); unit: Number of Prior Interventions] | 2.28 (2.75) | 2.26 (2.90) | 2.27 (2.82)

OUTCOME MEASURES:

1. Primary Outcome: Target Lesion Primary Patency at 6 Months
Description: Kaplan-Meier estimate of the time interval of uninterrupted patency from initial study treatment to the next access thrombosis or intervention performed on the target lesion.
  Six-month estimate of target lesion primary patency derived from Kaplan-Meier curve.
Time Frame: 6 months
Population: Percent of subjects maintaining patency based on Kaplan-Meier estimate based on per-protocol (effectiveness) population.
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | VIABAHN Treatment Group | PTA Treatment Group
Number analyzed (Participants) | 131 | 138
Percentage of Subjects | 52.9 [43.8 to 61.1] | 35.5 [27.4 to 43.6]

2. Primary Outcome: Target Lesion Primary Patency at 12 Months
Description: Kaplan-Meier estimate of the time interval of uninterrupted patency from initial study treatment to the next access thrombosis or intervention performed on the target lesion.
  Twelve-month estimate of target lesion primary patency derived from Kaplan-Meier curve.
Time Frame: 12 Months
Population: Percent of subjects maintaining patency based on Kaplan-Meier estimate based on per-protocol (effectiveness) population.
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | VIABAHN Treatment Group | PTA Treatment Group
Number analyzed (Participants) | 131 | 138
Percentage of Subjects | 30.2 [22.2 to 38.7] | 18.2 [12.1 to 25.2]

3. Secondary Outcome: Assisted Primary Patency at 6 Months
Description: Kaplan-Meier estimate of the time interval from initial study treatment to occlusion (thrombosis) of the vascular access circuit.
  Six-month estimate of assisted primary patency derived from Kaplan-Meier curve.
Time Frame: 6 months
Population: Percent of subjects maintaining patency based on Kaplan-Meier estimate based on per-protocol (effectiveness) population.
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | VIABAHN Treatment Group | PTA Treatment Group
Number analyzed (Participants) | 131 | 138
Percentage of Subjects | 56.2 [47.1 to 64.3] | 51.1 [42.3 to 59.2]
Statistical Analysis 1: Comparison: VIABAHN Treatment Group vs PTA Treatment Group; Test type: Superiority or Other; p = 0.530, Log Rank

4. Secondary Outcome: Assisted Primary Patency at 12 Months
Description: Kaplan-Meier estimate of the time interval from initial study treatment to occlusion (thrombosis) of the vascular access circuit.
  Twelve-month estimate of assisted primary patency derived from Kaplan-Meier curve.
Time Frame: 12 months
Population: Percent of subjects maintaining patency based on Kaplan-Meier estimate based on per-protocol (effectiveness) population.
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | VIABAHN Treatment Group | PTA Treatment Group
Number analyzed (Participants) | 131 | 138
Percentage of Subjects | 43.5 [34.5 to 52.1] | 35.3 [27.1 to 43.6]

5. Secondary Outcome: Assisted Primary Patency at 24 Months
Description: Kaplan-Meier estimate of the time interval from initial study treatment to occlusion (thrombosis) of the vascular access circuit.
  Twenty-four-month estimate of assisted primary patency derived from Kaplan-Meier curve.
Time Frame: 24 months
Population: Percent of subjects maintaining patency based on Kaplan-Meier estimate based on per-protocol (effectiveness) population.
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | VIABAHN Treatment Group | PTA Treatment Group
Number analyzed (Participants) | 131 | 138
Percentage of Subjects | 29.2 [21.0 to 38.0] | 29.0 [21.3 to 37.2]

6. Secondary Outcome: Access Secondary Patency at 6 Months
Description: Kaplan-Meier estimate of the time interval from initial study treatment to abandonment of the vascular access circuit.
  Six-month estimate of secondary access patency derived from Kaplan-Meier curve.
Time Frame: 6 months
Population: Percent of subjects maintaining patency based on Kaplan-Meier estimate based on per-protocol (effectiveness) population.
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | VIABAHN Treatment Group | PTA Treatment Group
Number analyzed (Participants) | 131 | 138
Percentage of Subjects | 91.2 [84.6 to 95.0] | 86.5 [79.5 to 91.3]
Statistical Analysis 1: Comparison: VIABAHN Treatment Group vs PTA Treatment Group; Test type: Superiority or Other; p = 0.475, Log Rank

7. Secondary Outcome: Access Secondary Patency [12 Months] Units Percentage of Subjects
Description: Kaplan-Meier estimate of the time interval from initial study treatment to abandonment of the vascular access circuit.
  Twelve-month estimate of secondary access secondary patency derived from Kaplan-Meier curve.
Time Frame: 12 months
Population: Percent of subjects maintaining patency based on Kaplan-Meier estimate based on per-protocol (effectiveness) population.
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | VIABAHN Treatment Group | PTA Treatment Group
Number analyzed (Participants) | 100 | 104
Percentage of Subjects | 82.7 [74.5 to 88.5] | 78.6 [70.3 to 84.8]

8. Secondary Outcome: Access Secondary Patency [24 Months] Units Percentage of Subjects
Description: Kaplan-Meier estimate of the time interval from initial study treatment to abandonment of the vascular access circuit.
  24-month estimate of secondary access secondary patency derived from Kaplan-Meier curve.
Time Frame: 24 months
Population: Percent of subjects maintaining patency based on Kaplan-Meier estimate based on per-protocol (effectiveness) population.
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | VIABAHN Treatment Group | PTA Treatment Group
Number analyzed (Participants) | 77 | 72
Percentage of Subjects | 68.9 [59.0 to 76.9] | 66.6 [57.1 to 74.6]

9. Primary Outcome: Target Lesion Primary Patency at 24 Months
Description: Kaplan-Meier estimate of the time interval of uninterrupted patency from initial study treatment to the next access thrombosis or intervention performed on the target lesion.
  P-Value calculated from 24-month data cohort after study completion.
Time Frame: 24 Months
Population: Percent of subjects maintaining patency based on Kaplan-Meier estimate based on per-protocol (effectiveness) population.
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | VIABAHN Treatment Group | PTA Treatment Group
Number analyzed (Participants) | 131 | 138
Percentage of Subjects | 15.7 [9.6 to 23.2] | 9.9 [5.5 to 15.9]
Statistical Analysis 1: Comparison: VIABAHN Treatment Group vs PTA Treatment Group; Test type: Superiority or Other; p = 0.008, Log Rank — P-value was calculated using Kaplan-Meier methodology with 24-month follow-up data

10. Primary Outcome: Freedom From Major Device, Procedure and Treatment Site-related Adverse Adverse Events Through 30 Days Post-procedure
Description: The primary safety endpoint is freedom from major device, procedure and treatment site-related adverse events through 30 days.
Time Frame: 30 days
Measure: Number; unit: Participants
Arm/Group | VIABAHN Treatment Group | PTA Treatment Group
Number analyzed (Participants) | 145 | 148
Participants | 0 | 2
Statistical Analysis 1: Comparison: VIABAHN Treatment Group vs PTA Treatment Group; Test type: Non-Inferiority or Equivalence — One-sided test of non-inferior proportions with delta = 0.15; p < 0.001, Z-test; One-sided

11. Secondary Outcome: Circuit Primary Patency
Description: Kaplan-Meier estimate of the time interval from initial study treatment to the next access thrombosis or intervention performed within the vascular access circuit.
  P-Value calculated from 24-month data cohort. Six-month estimate of circuit primary patency derived from Kaplan-Meier curve.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | VIABAHN Treatment Group | PTA Treatment Group
Number analyzed (Participants) | 145 | 148
Percentage of Subjects | 43.4 [34.6 to 51.9] | 29.4 [21.9 to 37.3]
Statistical Analysis 1: Comparison: VIABAHN Treatment Group vs PTA Treatment Group; Test type: Superiority or Other; p = 0.035, Log Rank

12. Secondary Outcome: Circuit Primary Patency [12 Months] Units Percentage of Subjects
Description: as for outcome 7
Time Frame: 12months
Population: Percent of subjects maintaining patency based on Kaplan-Meier estimate based on per-protocol (effectiveness) population.
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | VIABAHN Treatment Group | PTA Treatment Group
Number analyzed (Participants) | 48 | 38
Percentage of Subjects | 21.4 [14.4 to 29.3] | 15.2 [9.6 to 21.9]

13. Secondary Outcome: Circuit Primary Patency [24 Months] Units Percentage of Subjects
Description: as for outcome 7
Time Frame: 24 months
Population: Percent of subjects maintaining patency based on Kaplan-Meier estimate based on per-protocol (effectiveness) population.
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | VIABAHN Treatment Group | PTA Treatment Group
Number analyzed (Participants) | 12 | 9
Percentage of Subjects | 9.6 [4.9 to 16.1] | 6.8 [3.2 to 12.1]

14. Secondary Outcome: Clinical Success
Description: The resumption of normal dialysis for at least one session following study treatment (Index Procedure).
Time Frame: Following Index Procedure
Measure: Number; unit: Participants
Arm/Group | VIABAHN Treatment Group | PTA Treatment Group
Number analyzed (Participants) | 131 | 138
Participants
  Clinical Success = YES | 128 | 135
  Clinical Success = NO | 3 | 3
Statistical Analysis 1: Comparison: VIABAHN Treatment Group vs PTA Treatment Group; Test type: Superiority or Other; p = 1.000, Fisher Exact; Two-tailed

15. Secondary Outcome: Anatomic Success
Description: Less than 30 percent residual stenosis following study treatment (Index Procedure).
Time Frame: Index Procedure
Measure: Number; unit: Participants
Arm/Group | VIABAHN Treatment Group | PTA Treatment Group
Number analyzed (Participants) | 131 | 138
Participants
  Anatomic Success = YES | 131 | 116
  Anatomic Success = NO | 0 | 22
Statistical Analysis 1: Comparison: VIABAHN Treatment Group vs PTA Treatment Group; Test type: Superiority or Other; p < 0.001, Fisher Exact; Two-tailed

16. Secondary Outcome: Procedural Success
Description: Participants were considered to have Procedural Success if they achieved both anatomic success and clinical success.
Time Frame: Following Index Procedure
Measure: Number; unit: Participants
Arm/Group | VIABAHN Treatment Group | PTA Treatment Group
Number analyzed (Participants) | 131 | 138
Participants
  Procedural Success = YES | 128 | 113
  Procedural Success = NO | 3 | 25
Statistical Analysis 1: Comparison: VIABAHN Treatment Group vs PTA Treatment Group; Test type: Superiority or Other; p < 0.001, Fisher Exact; Two-tailed

ADVERSE EVENTS:
Arm/Group | VIABAHN Treatment Group | PTA Treatment Group
Serious Adverse Events (participants affected / at risk) | 78/145 | 77/148
Other Adverse Events (participants affected / at risk) | 4/145 | 8/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VIABAHN Treatment Group (N=145) | PTA Treatment Group (N=148)
Anemia (Blood and lymphatic system disorders) | 1 | 1
Anemia of chronic disease (Blood and lymphatic system disorders) | 1 | 0
Hypercoagulation (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Anginal pain (Cardiac disorders) | 3 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 2
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 4 | 2
Cardiac arrest (Cardiac disorders) | 6 | 8
Cardiopulmonary arrest (Cardiac disorders) | 3 | 2
Chest pain (Cardiac disorders) | 1 | 0
Congestive heart failure (Cardiac disorders) | 3 | 1
Coronary artery disease (Cardiac disorders) | 2 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 1 | 0
Junctional bradycardia (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 4 | 0
Non STEMI (Cardiac disorders) | 3 | 1
Tachycardia NOS (Cardiac disorders) | 1 | 0
Polycystic hepatorenal disease (Congenital, familial and genetic disorders) | 1 | 0
Addison's disease (Endocrine disorders) | 0 | 1
Blurry vision (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Retinal vascular occlusion (Eye disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abdominal pain aggravated (Gastrointestinal disorders) | 1 | 0
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 | 0
Acute duodenal ulcer with hemorrhage (Gastrointestinal disorders) | 0 | 1
Acute pancreatitis (Gastrointestinal disorders) | 0 | 1
Bleeding gastric ulcer (Gastrointestinal disorders) | 0 | 1
Blood in stool (Gastrointestinal disorders) | 2 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal hemorrhagic (Gastrointestinal disorders) | 0 | 1
GI bleed (Gastrointestinal disorders) | 3 | 2
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastroparesis (Gastrointestinal disorders) | 1 | 0
Hematochezia (Gastrointestinal disorders) | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0
Internal hemorrhoids (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal bleeding (Gastrointestinal disorders) | 1 | 0
Melena (Gastrointestinal disorders) | 0 | 1
Mesenteric ischemia (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute on chronic (Gastrointestinal disorders) | 1 | 0
Pancreatitis due to gallstones (Gastrointestinal disorders) | 0 | 1
Peptic ulcer disease (Gastrointestinal disorders) | 1 | 0
Rectal bleeding (Gastrointestinal disorders) | 1 | 0
Right-sided colitis (Gastrointestinal disorders) | 1 | 0
Small bowel obstruction (Gastrointestinal disorders) | 2 | 1
Upper gastrointestinal bleeding (Gastrointestinal disorders) | 2 | 2
Upper gastrointestinal symptoms (Gastrointestinal disorders) | 2 | 0
Adverse drug reaction (General disorders) | 0 | 1
Catheter site bleeding (General disorders) | 1 | 0
Chest pain (General disorders) | 8 | 6
Debility marked (General disorders) | 0 | 1
Ill-defined disorder (General disorders) | 0 | 1
Incarcerated hernia (General disorders) | 0 | 1
Intraocular lens dislocation (General disorders) | 0 | 1
Pain at rest (General disorders) | 0 | 1
Peritoneal catheter dysfunction (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 1 | 0
Acute cholecystitis (Hepatobiliary disorders) | 1 | 0
Biliary stasis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 1
Allergic reaction to antibiotics (Immune system disorders) | 1 | 2
Abscess dental (Infections and infestations) | 0 | 1
Abscess leg (Infections and infestations) | 1 | 0
Abscess of finger (Infections and infestations) | 1 | 0
Acute tracheobronchitis (Infections and infestations) | 1 | 0
Arteriovenous graft site infection (Infections and infestations) | 5 | 9
Bacteremia (Infections and infestations) | 5 | 0
Bacterial endocarditis (Infections and infestations) | 1 | 0
Biliary sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 3 | 0
C.difficile colitis (Infections and infestations) | 2 | 0
Candida sepsis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 2 | 0
Cellulitis of arm (Infections and infestations) | 0 | 1
Cellulitis of foot (Infections and infestations) | 1 | 0
Cellulitis of leg (Infections and infestations) | 2 | 0
Cellulitis of legs (Infections and infestations) | 0 | 1
Community acquired pneumonia (Infections and infestations) | 2 | 1
Diabetic foot infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Foot infection (Infections and infestations) | 2 | 0
Gangrene (Infections and infestations) | 5 | 5
Hospital acquired infection (Infections and infestations) | 1 | 0
Infection of amputation stump (Infections and infestations) | 1 | 0
Leg infection (Infections and infestations) | 1 | 1
Osteomyelitis (Infections and infestations) | 3 | 1
Pneumonia (Infections and infestations) | 2 | 8
Pneumonia aspergillus (Infections and infestations) | 0 | 1
Recurrent urinary tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 5 | 5
Sepsis MRSA (Infections and infestations) | 1 | 2
Septic shock (Infections and infestations) | 3 | 0
Shingles (Infections and infestations) | 0 | 1
Staphylococcal bacteremia (Infections and infestations) | 2 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 2
Streptococcal cellulitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 4
Urosepsis (Infections and infestations) | 1 | 0
Viral syndrome (Infections and infestations) | 0 | 1
Acute subdural hematoma (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 1
Arteriovenous graft aneurysm (Injury, poisoning and procedural complications) | 1 | 1
Arteriovenous graft site bleeding (Injury, poisoning and procedural complications) | 4 | 3
Arteriovenous graft site hematoma (Injury, poisoning and procedural complications) | 0 | 2
Arteriovenous graft site hemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Bleeding postoperative (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture C2 (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fat embolism (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture of upper end or unspecified part of tibia and fibula, closed (Injury, poisoning and procedural complications) | 1 | 0
Hemodialysis-induced symptom (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Hypotension during dialysis (Injury, poisoning and procedural complications) | 0 | 2
Lower limb wound (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 2
Postoperative bleeding (Injury, poisoning and procedural complications) | 0 | 1
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 | 1
Pubic rami fracture (Injury, poisoning and procedural complications) | 1 | 0
Electrocardiogram abnormal non-specific (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 0
Diabetes mellitus poor control (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 5 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 6 | 7
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 3
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Volume overload (Metabolism and nutrition disorders) | 11 | 5
Avascular necrosis femoral head (Musculoskeletal and connective tissue disorders) | 1 | 0
Hand pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Jaw pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Leg pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis aggravated (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis of cervical spine (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in arm (Musculoskeletal and connective tissue disorders) | 1 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 4
Dizziness (Nervous system disorders) | 1 | 0
Encephalopathy acute (Nervous system disorders) | 0 | 2
Slurred speech (Nervous system disorders) | 1 | 0
Stroke (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 1
Tonic-clonic seizures (Nervous system disorders) | 0 | 1
Toxic encephalopathy (Nervous system disorders) | 0 | 1
Transient ischemic attack (Nervous system disorders) | 2 | 1
Tremor (Nervous system disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 3 | 2
End stage renal disease (ESRD) (Renal and urinary disorders) | 2 | 4
Hematuria (Renal and urinary disorders) | 0 | 1
Kidney failure (Renal and urinary disorders) | 1 | 0
Renal mass (Renal and urinary disorders) | 0 | 2
Uremia (Renal and urinary disorders) | 0 | 2
Acute on chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Flash pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung nodule (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Non-cardiogenic pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Orthopnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Vocal cord dysfunction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Facial swelling (Skin and subcutaneous tissue disorders) | 1 | 0
Foot ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Heel ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Leg ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Venous stasis ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Anticoagulant therapy (Surgical and medical procedures) | 1 | 0
Blood pressure management (Surgical and medical procedures) | 1 | 0
Kidney transplant (Surgical and medical procedures) | 1 | 0
Toe amputation (Surgical and medical procedures) | 0 | 1
Accelerated Hypertension (Vascular disorders) | 1 | 0
Arterial embolism NOS (Vascular disorders) | 0 | 1
Atherosclerosis of arteries of the extremities (Vascular disorders) | 1 | 0
Critical limb ischemia (Vascular disorders) | 1 | 0
Deep venous thrombosis arm (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Hypertensive emergency (Vascular disorders) | 0 | 1
Hypertensive urgency (Vascular disorders) | 1 | 2
Malignant hypertension (Vascular disorders) | 1 | 1
Peripheral arterial disease (Vascular disorders) | 1 | 2
Peripheral ischemia (Vascular disorders) | 0 | 2
Uncontrolled hypertension (Vascular disorders) | 1 | 0
Venous (peripheral) insufficiency, unspecified (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VIABAHN Treatment Group (N=145) | PTA Treatment Group (N=148)
Chest pain (General disorders) | 4 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No